CLINICAL TRIAL: NCT01307969
Title: Formulations of Liposomal Local Anesthetics for Dental Anesthesia
Brief Title: Formulations of Liposomal Local Anesthetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Michelle Franz-Montan, Unicamp
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 164/2006
Record Dates: First submitted 2011-02-16; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-02

CONDITIONS: Underdosing of Local Anesthetics, Initial Encounter
Keywords: liposomes; ropivacaine; dental anesthesia; dentistry
MeSH Terms: interventions — Ropivacaine; Liposomes; Epinephrine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anesthetic efficacy (Experimental): Local anesthetics were injected at the apex of the maxillary right canine.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 1,8 mL of the local anesthetic formulations were injected at the apex of the maxillary right canine.
  Other Names: 0,5% ropivacaine encapsulated in liposomes; 0,5% ropivacaine with epinephrine 1:200.000; 2% lidocaine with epinephrine 1:100.000

SUMMARY:
This blinded cross-over study aim to evaluate the efficacy of liposome-encapsulated ropivacaine formulation for dental anesthesia.

DETAILED DESCRIPTION:
This blinded cross-over study aim to evaluate the efficacy of liposome-encapsulated 0, 5% ropivacaine for dental anesthesia after maxillary infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Volunteers were free from cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and haematological diseases, psychiatric disorders and allergy to local anesthetics

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
After anesthetic injection the pulpal response was assessed by an electrical pulp tester. | 100 minutes

SECONDARY OUTCOMES:
Duration of soft tissue anesthesia was measured as the time from beginning to end of lip and gingival numbness. | 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Franz-Montan, PhD, Principal Investigator — Researcher at Unicamp
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Derived] Franz-Montan M, de Paula E, Groppo FC, Ranali J, Volpato MC. Efficacy of liposome-encapsulated 0.5% ropivacaine in maxillary dental anaesthesia. Br J Oral Maxillofac Surg. 2012 Jul;50(5):454-8. doi: 10.1016/j.bjoms.2011.07.010. Epub 2011 Aug 9. PMID 21831487